CLINICAL TRIAL: NCT04068142
Title: The Acceptability and Feasibility of an ED-based, Peer-delivered, Suicide Safety Planning Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 239486
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-10

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Mental Health Issue
Keywords: Suicide; Suicide Prevention; Safety Planning
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Personnel Safety Planning (No Intervention): Patients will complete a traditional written suicide safety plan with clinical personnel.
- Peer Supporter Safety Planning (Experimental): Patients will complete a traditional written suicide safety plan with peer supporters.
  Interventions: Other: Peer Supporter Safety Planning

INTERVENTIONS:
Other: Peer Supporter Safety Planning — The rationale for testing a peer-delivered intervention in the ED relies on the following evidence: a) a peer is an individual with lived experience who is now supporting other mental health patients in crisis; b) the experience of a mental health patient in the ED often shapes the perception of the health system, and may influence willingness to seek future care; c) peers may provide more empathetic care than providers without lived experience, which may positively impact patients; d) peer-based programs for patients with serious mental illness that do not involve safety planning are at least as good as non-peer based programs at preventing hospitalizations and promoting engagement in care, with the most promising interventions involving self-management or peer-navigator roles; and e) existing evidence from high-quality studies is scarce, but in moderate-low quality studies has indicated that peers are no less effective than mental health workers
  Arms: Peer Supporter Safety Planning

SUMMARY:
Safety planning is a brief, ED-feasible intervention which has been demonstrated to save lives, and has been universally recommended by every recent expert consensus panel on suicide prevention strategies. In one popular version of the safety plan developed by Stanley et al, the patient is encouraged to write out the following items: identifying personal signs of a crisis; helpful internal coping strategies; social contacts or settings which may distract from a crisis; using family members or friends for help when in crisis; mental health professionals who can be contacted when in crisis; and restricting access to lethal means. In most emergency departments, safety-planning is done by clinical personnel such as psychologists or social workers, but these providers are often too busy to perform safety-planning well or have multiple other patient care responsibilities.

This study aims to find out if ED patients prefer to complete a safety plan with a peer supporter or clinical personnel. People who are visiting the emergency department for thoughts of self-harm will be asked to participate.

DETAILED DESCRIPTION:
This project aims to answer the following three research questions: (1) In general, do ED patients with suicidal ideation/attempt prefer to interact with/receive support from peers with life experiences of suicide or clinical professionals who might have such life experiences or not? (2) Will patients with suicidal ideation/attempt accept a peer-delivered safety planning intervention as opposed to one delivered by clinical personnel? (3) Are peer-delivered safety plans of equal quality as those delivered by clinical personnel?

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for suicidal ideation (SI) or after a suicide attempt to the University of Arkansas for Medical Sciences (UAMS) Emergency Department (ED)
* Willingness to engage in safety planning with trained non-clinical staff
* English-speaking and English-writing (as translators will not be available for this study)

Exclusion Criteria:

* <18 or >89 years of age
* Patients appearing critically-ill
* Incarcerated or in police custody
* Currently intoxicated with alcohol or other substance
* ED staff objection to patient enrollment in study
* Unwilling or unable to complete the safety plan with a peer supporter
* Unwilling or unable to show the safety plan to clinical staff

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Wilson, M.D., Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson MP, Waliski A, Thompson RG Jr. Feasibility of Peer-Delivered Suicide Safety Planning in the Emergency Department: Results From a Pilot Trial. Psychiatr Serv. 2022 Oct 1;73(10):1087-1093. doi: 10.1176/appi.ps.202100561. Epub 2022 May 3. PMID 35502515

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer Supporter Safety Planning: Patients will complete a traditional written suicide safety plan with peer supporters.
  Peer Supporter Safety Planning: The rationale for testing a peer-delivered intervention in the emergency department (ED) relies on the following evidence: a) a peer is an individual with lived experience who is now supporting other mental health patients in crisis; b) the experience of a mental health patient in the ED often shapes the perception of the health system, and may influence willingness to seek future care; c) peers may provide more empathetic care than providers without lived experience, which may positively impact patients; d) peer-based programs for patients with serious mental illness that do not involve safety planning are at least as good as non-peer based programs at preventing hospitalizations and promoting engagement in care, with the most promising interventions involving self-management or peer-navigator roles; and e) existing evidence from high-quality studies is scarce, but in moderate-low quality studies has indicated that peers are no less effective than mental health workers
Period: Overall Study
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning
Started | 17 | 20
Completed | 15 | 16
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45 [34 to 54.5] | 38.5 [28.5 to 42.8] | 39 [29 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Suicidal Ideology (SI) Participants Who Agree to Receive a Safety Plan
Description: Evaluate the number of suicidal ideology (SI) patients approached in the ED who agree to receive a safety plan.
Time Frame: approach in the ED (typically <1 hour)
Population: participants
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning
Number analyzed (Participants) | 15 | 16
Participants | 15 | 16

2. Primary Outcome: Proportion of Eligible Patients
Description: Evaluate the proportion of patients approached who meet all inclusion/exclusion criteria.
Time Frame: Up to 12 hours
Population: participants
Measure: Count of Participants; unit: Participants
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning
Number analyzed (Participants) | 17 | 20
Participants | 17 | 20

3. Primary Outcome: Quality of Safety Plans
Description: Evaluate the quality of the completed safety plans. This will be done by retrospective review after the patient has left the ED. Safety plans will be graded individually, then resolved by consensus, for quality (0=blank, 1=boilerplate, 2=some evidence of personalization, 3=highly personalized; range=0-24) by the investigators using materials developed by Brown and Stanley for this purpose. Using a "safety checklist," responses for each of the 6 safety plan steps will be classified according to the personalization of the information in each step.
Time Frame: Up to 12 hours
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning
Number analyzed (Participants) | 15 | 16
scores on a scale | 8 [7 to 9] | 12.5 [10 to 16.5]

4. Primary Outcome: Satisfaction With Safety Planning
Description: Evaluate patient satisfaction with safety planning. This will be assessed by having the patient rate their experience with the safety planning process on a 7-point Likert scale (1 - strongly disagree; 2 - disagree; 3 - moderately disagree; 4 - neutral; 5 - moderately agree; 6 - agree; 7 - strongly agree). A Likert scale measures how much someone disagrees or agrees with a particular statement.
Time Frame: Up to 12 hours
Population: participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning
Number analyzed (Participants) | 15 | 16
score on a scale | 4 [4 to 4] | 4.5 [4 to 6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while safety planning (typically 1 hour or less). Mortality was assessed in the medical record 30 days after ED discharge.
Arm/Group | Clinical Personnel Safety Planning | Peer Supporter Safety Planning
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT04068142/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT04068142/ICF_001.pdf